CLINICAL TRIAL: NCT05716867
Title: The Evidence of Early Childhood Caries Prediction by Salivary Cystatin S Levels in a Group of Egyptian Children: a Case Control Study
Brief Title: Salivary Cystatin S Levels in a Group of Egyptian Children
Status: Active, not recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tasneem Salah Sayed Mohamed Abo Ali, principle investigator, Cairo University
Other Study IDs: PEDO 1-2-1
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Early Childhood Caries
Keywords: early childhood caries, salivary cystatin S protein, salivary buffer capacity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Children with early childhood caries aged between 36-71 month
  Interventions: Biological: Measurement of salivary cystatin S protein levels in saliva
- Caries free children aged between 36-71 month
  Interventions: Biological: Measurement of salivary cystatin S protein levels in saliva

INTERVENTIONS:
Biological: Measurement of salivary cystatin S protein levels in saliva — The human cystatin S enzyme-linked immunosorbent assay (ELISA) kit will be used to measure the amounts of cystatin S in saliva for cases and controls

SUMMARY:
Aim of the study

1. Measuring the levels of salivary cystatin S protein and salivary buffering capacity to determine their relation to early childhood caries.
2. Predection of early childhood caries by using salivary cystatin S levels with demographic, clinical and nutrition habits characteristics of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Medically free children aged 36 to 71 months with one or more decayed (noncavitated or cavitated lesions), missing, or filled teeth due to caries in any primary tooth(cases).
* Medically free children aged 36 to 71 months with no decayed, missing, or filled teeth due to caries in any primary tooth(controls).

Exclusion Criteria:

* Children receiving antibiotic therapy within three month and fluoride prophylaxis within one year.
* Parents who will refuse to participate or refuse to sign the informed consent.
* Children who will not agree or cooperate with participation.

Ages: 36 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: the patients going to diagnosis clinic of Pediatric dentistry and Dental Public Health Department, Cairo University
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Levels of salivary cystatin S protein | 2 months
  Levels of salivary cystatin S protein measured by Human cystatin S enzyme linked immunosorbent assay (ELISA) kit (unit ng/ml)

SECONDARY OUTCOMES:
Buffer Capacity | 2 months
  Buffer Capacity measured by PH meter
Demographic, clinical and nutrition habits characteristics of participants Interview | 2 months
  Demographic, clinical and nutrition habits characteristics of participants, using interview

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided